CLINICAL TRIAL: NCT07166874
Title: The Impacts of Gluten Free Diet on Disease Activity, Quality of Life and Intestinal Permeability in Patients Diagnosed With Ankylosing Spondylitis.
Brief Title: The Impacts of Gluten-free Diet in Patients With Ankylosing Spondylitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Gülay Sezgin, Dietitian, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20240704
Record Dates: First submitted 2025-08-26; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Ankylosing Spondylitis
Keywords: gluten free diet; intestinal permeability; zonulin; ankylosing spondylitis; cytokine; BASDAI
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — Diet, Gluten-Free

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): In the control arm, patients will continue their eating habits.
- Gluten Free Diet (Experimental): Patients in the experimental arm will received a gluten-free diet for 8 weeks.
  Interventions: Behavioral: Gluten Free Diet

INTERVENTIONS:
Behavioral: Gluten Free Diet — Patients in the experimental arm will received a gluten-free diet for 8 weeks.
  Arms: Gluten Free Diet

SUMMARY:
Subclinical intestinal inflammation and intestinal permeability have been reported in patients with ankylosing spondylitis. Gluten is one of the main triggers of zonulin releaseand gluten intake may contribute to the development of the disease by increasing intestinal permeability. This study aims to determine the impacts of a gluten-freediet on intestinal permeability, sub-clinical intestinal inflammation, disease activity, functional status and quality of life in patients with ankylosing spondylitis. The main questions it aims to answer are:

Does a gluten-free diet have an effect on disease activity and functional status in patients with ankylosing spondylitis? Does a gluten-free diet have an effect on intestinal permeability and subclinical intestinal inflammation in patients with ankylosing spondylitis? The investigators will evaluate the effects of the gluten-free diet compared to a control group.

DETAILED DESCRIPTION:
Ankylosing Spondylitis (AS) is a chronic, progressive, inflammatory rheumatic disease that severely impairs patients' quality of life and functional capacity. The gut-joint axis theory in the pathogenesis of AS is gaining increasing support. Specifically, the increase in intestinal permeability mediated by zonulin, and the subsequent leakage of bacterial products (e.g., LPS) into the circulation, is recognized as a central mechanism in many diseases, including AS. Gluten has been proven to be one of the most potent dietary triggers of zonulin release, independent of genetic predisposition. Despite this, the clinical effects of a gluten-free diet (GFD) on this specific mechanism and its potential in AS patients have not yet been fully elucidated. Although indirect evidence suggesting that a GFD may provide clinical improvement in AS patients is accumulating, there are no studies in the literature that directly test the underlying biological mechanism (zonulin → LPS → systemic inflammation). This represents a critical knowledge gap that prevents clinicians from providing evidence-based dietary recommendations to patients. Therefore, investigators basically propose two hypotheses.

Hypothesis 1: An 8-week gluten-free diet in patients with Ankylosing Spondylitis will improve intestinal barrier integrity by reducing gliadin-induced zonulin release.

Hypothesis 2: The reduction in intestinal permeability will decrease the amount of lipopolysaccharide (LPS) translocating into the circulation and the subsequent pro-inflammatory cytokine response (TNF-α, IL-6). Consequently, this mechanism will lead to a measurable clinical improvement in disease activity (BASDAI) and quality of life (ASQoL).

To this end, an 8-week, randomized controlled prospective intervention study has been designed, which will include 60 AS patients aged 18-64. The intervention group (Gluten-Free Diet Group, n=30) will follow a gluten-free diet for 8 weeks in addition to their current treatments. The daily energy requirement for patients in this group will be calculated (using the Harris-Benedict equation for basal metabolic rate, adjusted for physical activity levels), and a gluten-free diet will be planned accordingly. In the initial face-to-face meeting, a dietitian will explain how to properly adhere to participants the gluten-free diet.Compliance will be monitored by the dietitian at weeks 2, 4, and 6 using a 1-day food record. Patients who do not adhere to the gluten-free diet will be excluded from the study. The control group (n=30) will continue with their current standard clinical follow-up without any dietary intervention. Disease activity, functional status, gastrointestinal symptoms, and quality of life will be assessed using the Bath Ankylosing Spondylitis Disease Activity Index (BASDAI), the Bath Ankylosing Spondylitis Functional Index (BASFI), the Gastrointestinal Symptom Rating Scale (GSRS), and the Ankylosing Spondylitis Quality of Life (ASQoL) questionnaire. All biochemical measurements will be performed at baseline and at the end of the 8th week. This design will allow us to evaluate whether a GFD provides an additional benefit to standard care in real-world clinical practice.

The primary objective of the study is to measure the effect of a GFD on markers of intestinal permeability (serum zonulin) and microbial translocation (serum LPS). The secondary objectives are to evaluate the reflections of this mechanistic change on systemic inflammation markers (CRP, TNF-α, IL-6) and clinical disease activity scores (BASDAI, ASQoL). Measurements will be performed using validated ELISA methods and standard clinical questionnaires.

The primary novelty of this project is that it will be one of the first studies to explain the efficacy of a GFD in AS patients by targeting the underlying biological mechanism (zonulin → LPS → inflammation). The findings obtained at the end of the project will contribute to the development of evidence-based dietary recommendations for the management of AS.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of axial SpA defined by ASAS criteria
* Adults (aged 18-64 years)
* stable treatment (NSAID and/or DMARD) for at least 3 months
* provide written informed consent and submit to the requirements of the study

Exclusion Criteria:

* Any diet at the time of inclusion or within 3 months prior to inclusion;
* have a history of celiac disease;
* have a history of Ulcerative Colitis, Crohn's Disease and Irritable Bowel Syndrom
* patients with Type 1 and Type 2 Diabetes Mellitus
* patients with Hashimoto Thyroiditis
* are pregnant, breastfeeding,
* patients who have used omega-3 and vitamins (A, C, E) regularly in the last 3 months.
* BMI <18,50 kg/m2
* BMI ≥29,99 kg/m2

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-31 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
effects of a 8-week Gluten Free Diet versus placebo diet on fasting serum zonulin levels | Change from baseline serum zonulin at 8 weeks
  Serum zonulin will be evaluated as a biomarker of intestinal permeability. It will be measured by ELISA(enzyme-linked immunosorbent assay) method.
effects of a 8-week Gluten Free Diet versus placebo diet on fasting serum LPS levels | Change from baseline serum LPS at 8 weeks
  Serum LPS will be evaluated as a biomarker of intestinal permeability. It will be measured by ELISA(enzyme-linked immunosorbent assay) method.

SECONDARY OUTCOMES:
effects of a 8 week Gluten Free Diet versus placebo diet on the activity of Ankylosing Spondylitis evaluated by the Bath Ankylosing Spondylitis Disease Activity Index (BASDAI). | Change from baseline BASDAI score at 8 weeks
  The BASDAI consists of a 0 - 10 scale measuring discomfort, pain, and fatigue (0 being no problem and 10 being the worst problem) in response to six questions. The resulting 0 to 50 score is divided by 5 to give a final 0 - 10 BASDAI score. Scores of 4 or greater suggest suboptimal control of disease,
effects of a 8-week Gluten Free Diet versus placebo diet on functional disability asssessed by Bath Ankylosing Spondylitis Functionnal Index (BASFI) questionnaire | Change from baseline BASFI score at 8 weeks
  Functional disability index consisting of 10 questions. After taking the answer of each question out of 10, the total of the points was calculated by dividing the number of questions. The higher the score, the greater the handicap.
effects of a 8 week Gluten Free Diet versus placebo diet on the quality of life of Ankylosing Spondylitis evaluated by the Ankylosing Spondylitis Quality of Life Questionnaire (ASQoL). | Change from baseline ASQoL score at 8 weeks
  It evaluates quality of life. Each statement on the ASQoL (18-item) is given a score of "1" or "0".
  A score of "1" is given where the item is affirmed, indicating adverse QoL. All item scores are summed to give a total score or index. Scores can range from 0 (good QoL) to 18 (poor QoL).
effects of a 8-week Gluten Free Diet versus placebo diet on CRP levels | Change from baseline CRP at 8 weeks
  A c-reactive protein test measures the level of c-reactive protein (CRP) in your blood. CRP is a protein made by your liver. It's sent into your bloodstream in response to inflammation. Normally, you have low levels of c-reactive protein in your blood. High levels may be sign of a serious infection or other disorder.
effects of a 8-week Gluten Free Diet versus placebo diet on ESR levels | Change from baseline ESR at 8 weeks
  An ESR is a type of blood test that measures how quickly erythrocytes settle at the bottom of a test tube that contains a blood sample. Normally, red blood cells settle relatively slowly. A faster-than-normal rate may indicate inflammation in the body.
effects of a 8 week gluten free diet versus placebo diet on the gastrointestinal symptoms | Change from baseline GSRS score at 8 weeks
  Validated seven point questionnaire that assesses gastrointestinal symptoms for five symptom areas, including abdominal pain, reflux, indigestion, diarrhea, and constipation. Individual scores are calculated for each symptom area and the mean of the scores is used to derive an overall GSRS score. Scores range from 0-7, with higher scores indicating gastrointestinal discomfort.
change in body weight | Change from baseline body weight at 8 weeks
  Body weight will be measured with a bathroom scale.
change in Body Mass Index | Change from baseline BMI at 8 weeks
  The BMI will be calculated by the formula (height/weight²).
effects of a 8-week Gluten Free Diet versus placebo diet on fasting glucose levels | Change from baseline fasting glucose at 8 weeks
  Glucose level testing will be done after an overnight fast.
effects of a 8-week Gluten Free Diet versus placebo diet on fasting insulin levels | Change from baseline fasting insulin at 8 weeks
  Insuline level testing will be done after an overnight fast.
effects of a 8-week Gluten Free Diet versus placebo diet on fasting serum calprotectin levels | Change from baseline serum calprotektin at 8 weeks
  Serum calprotectin will be evaluated as a biomarker of subclinical intestinal inflammation. It will be measured by ELISA(enzyme-linked immunosorbent assay) method.
effects of a 8-week Gluten Free Diet versus placebo diet on fasting serum haptoglobin levels | Change from baseline serum haptoglobin at 8 weeks
  Haptoglobin is an acute phase reactant. Serum haptoglobin will be evaluated as a biomarker of inflammation. It will be measured by ELISA(enzyme-linked immunosorbent assay) method.
effects of a 8-week Gluten Free Diet versus placebo diet on fasting serum TNF-alpha levels | Change from baseline serum TNF-alpha at 8 weeks
  Serum TNF-alpha will be evaluated as a biomarker of inflammation. It will be measured by ELISA(enzyme-linked immunosorbent assay) method.
effects of a 8-week Gluten Free Diet versus placebo diet on fasting serum IL-6 levels | Change from baseline serum IL-6 at 8 weeks
  Serum IL-6 will be evaluated as a biomarker of inflammation. It will be measured by ELISA(enzyme-linked immunosorbent assay) method.
effects of a 8-week Gluten Free Diet versus placebo diet on fasting serum IL-10 levels | Change from baseline serum IL-10 at 8 weeks
  Serum IL-10 will be evaluated as a biomarker of inflammation. It will be measured by ELISA(enzyme-linked immunosorbent assay) method.

CONTACTS AND LOCATIONS:
Locations (4):
- Turkey (Türkiye) (4):
  - Bakırköy Dr. Sadi Konuk Training and Research hospital, Istanbul
  - İstanbul Medeniyet University, Istanbul
  - İstanbul Sağlık Bilimleri University, Istanbul
  - Marmara University, Istanbul

IPD SHARING:
Plan to Share IPD: No